CLINICAL TRIAL: NCT05329649
Title: A Phase 3 Study to Evaluate the Safety and Efficacy of a Single Dose of CTX001 in Pediatric Subjects With Severe Sickle Cell Disease
Brief Title: Evaluation of Safety and Efficacy of CTX001 in Pediatric Participants With Severe Sickle Cell Disease (SCD)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Collaborators: CRISPR Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX21-CTX001-151; 2021-002173-26 (EudraCT Number)
Record Dates: First submitted 2022-04-07; First posted 2022-04-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Sickle Cell Disease; Hydroxyurea Failure; Hydroxyurea Intolerance; Hemoglobinopathies; Hematological Diseases
MeSH Terms: conditions — Anemia, Sickle Cell; Hemoglobinopathies; Hematologic Diseases | interventions — exagamglogene autotemcel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CTX001 (Experimental): CTX001 (autologous CD34+ hHSPCs modified with CRISPR-Cas9 at the erythroid lineage-specific enhancer of the BCL11A gene). Participants will receive single infusion of CTX001 through central venous catheter.
  Interventions: Biological: CTX001

INTERVENTIONS:
Biological: CTX001 — Administered by intravenous infusion following myeloablative conditioning with busulfan.
  Other Names: Exagamglogene autotemcel; Exa-cel

SUMMARY:
This is a single-dose, open-label study in pediatric participants with severe SCD and hydroxyurea (HU) failure or intolerance. The study will evaluate the safety and efficacy of autologous CRISPR-Cas9 modified CD34+ human hematopoietic stem and progenitor cells (hHSPCs) (CTX001).

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of severe SCD as defined by:
* Documented SCD genotypes
* History of at least two severe VOCs events per year for the previous two years prior to enrollment
* Hydroxyurea (HU) failure unless HU intolerant
* Eligible for autologous stem cell transplant as per investigators judgment

Key Exclusion Criteria:

* A willing and healthy 10/10 human leukocyte antigen (HLA)-matched related donor
* Prior hematopoietic stem cell transplant (HSCT).
* Clinically significant and active bacterial, viral, fungal, or parasitic infection

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2022-05-02 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants who do not Have any Severe Vaso-occlusive Crises (VOCs) for at Least 12 Consecutive Months (VF12) | Up to 24 Months After CTX001 Infusion

SECONDARY OUTCOMES:
Proportion of Participants Free from Inpatient Hospitalization for Severe VOCs for at Least 12 Months (HF12) | Up to 24 Months After CTX001 Infusion
Relative Reduction in Annualized Rate of Severe VOCs | From Baseline up to 24 Months After CTX001 Infusion
Duration of Severe VOC Free in Participants who Have Achieved VF12 | Up to 24 Months After CTX001 Infusion
Relative Reduction in Annualized Rate of Inpatient Hospitalizations for Severe VOCs | From Baseline up to 24 Months After CTX001 Infusion
Proportion of Participants With Sustained Fetal Hemoglobin (HbF) ≥20 Percent (%) for at Least 3 Months | Up to 24 Months After CTX001 Infusion
Proportion of Participants With Sustained HbF ≥20% for at Least 6 Months | Up to 24 Months After CTX001 Infusion
Proportion of Participants With Sustained HbF ≥20% for at Least 12 Months | Up to 24 Months After CTX001 Infusion
Proportion of Alleles With Intended Genetic Modification Present in Peripheral Blood Over Time | Up to 24 Months After CTX001 Infusion
Proportion of Alleles With Intended Genetic Modification Present in CD34+ Cells of the Bone Marrow Over Time | Up to 24 Months After CTX001 Infusion
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Signing of Informed Consent up to 24 Months After CTX001 Infusion
Proportion of Participants With Engraftment (First day of 3 Consecutive Measurements of Absolute Neutrophil Count [ANC] ≥500 per Microliter [mcgL] on 3 Different Days) | Within 42 Days After CTX001 Infusion
Time to Engraftment | Up to 24 Months After CTX001 Infusion
Incidence of Transplant-related Mortality (TRM) Within 100 Days After CTX001 Infusion | Within 100 Days After CTX001 infusion
Incidence of TRM Within 12 Months After CTX001 Infusion | Within 12 Months After Infusion
Incidence of All-cause Mortality | From Signing of Informed Consent up to 24 Months After CTX001 Infusion
Relative Reduction in Annualized Duration of Hospitalization for Severe VOCs | From Baseline up to 24 Months After CTX001 Infusion
Proportion of Participants With Sustained HbF ≥30% for at Least 3 Months | Up to 24 Months After CTX001 Infusion
Proportion of Participants With Sustained HbF ≥30% for at Least 6 Months | Up to 24 Months After CTX001 Infusion
Proportion of Participants With Sustained HbF ≥30% for at Least 12 Months | Up to 24 Months After CTX001 Infusion
Time for Participants to Reach HbF ≥20% | Up to 24 Months After CTX001 Infusion
Time for Participants to Reach HbF ≥30% | Up to 24 Months After CTX001 Infusion
Relative Reduction from Baseline in Annualized Volume and Episodes of RBC Transfusions for SCD-related indications starting after Month 12 post-CTX001 infusion | Up to 24 Months After CTX001 Infusion
HbF Concentrations Over Time | Up to 24 Months After CTX001 Infusion
Hemoglobin (Hb) Concentrations Over Time | Up to 24 Months After CTX001 Infusion
Change in Reticulocyte Count Over Time | From Baseline up to 24 Months After CTX001 Infusion
Change in Indirect Bilirubin Over Time | From Baseline up to 24 Months After CTX001 Infusion
Change in Haptoglobin Over Time | From Baseline up to 24 Months After CTX001 Infusion
Proportion of Participants with Detectable Haptoglobin Over Time | Up to 24 Months After CTX001 Infusion
Change in Lactate Dehydrogenase (LDH) Over Time | From Baseline (Pre-infusion) up to 24 Months After CTX001 Infusion
Proportion of Participants with Normalized LDH Over Time | Up to 24 Months After CTX001 Infusion

CONTACTS AND LOCATIONS:
Locations (7):
- United States (4):
  - Levine Children's Hospital - Hematology, Charlotte, North Carolina
  - The Children's Hospital of Philadelphia - Hematology, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - TriStar Medical Group Children's Specialists - Pediatric Oncology, Nashville, Tennessee
- University Hospital Duesseldorf - Department of Pediatric Oncology, Hematology and Clinical Immunology, Düsseldorf, Germany
- IRCSS Ospedale Pediatrico Bambino Gesu - Dipartimento di Onco-Ematologia e Terapia Cellulare e Genica, Rome, Italy
- St.Mary's Hospital - Haematology Dept, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing